CLINICAL TRIAL: NCT01913808
Title: Efficacy of Intravenous Ferric Carboxymaltose in the Improvement of Anemia in Patients With Postoperative Knee Prosthesis
Brief Title: Comparing Intravenous and Oral Iron in Postoperative Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Principal Investigator, Elvira Bisbe, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEV-POST/ESP10; 2010-023038-22 (EudraCT Number)
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Anemia; Osteoarthritis, Knee
Keywords: Postoperative anemia; Total knee arthroplasty; Iron therapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — ferric carboxymaltose; ferroglycine sulfate; Iron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric carboxymaltose (Experimental): Ferric carboxymaltose (Ferinject®, Vifor-France) was given as a single i.v. dose to correct the total iron deficit calculated by the Ganzoni formula (total iron deficit [mg] = 2.4 x patient's weight [kg] x (target Hb [13 g/dL] - current Hb [g/dL]) + 500 [mg iron stores]
  Interventions: Drug: Ferric carboxymaltose
- Ferrous glycine sulphate (Active Comparator): Ferrous glycine sulphate (Ferbisol-Bial Industrial Farmacéutica, Spain) was given as a once daily oral dose of 100 mg iron from the day of discharge (Day 7) to the rehabilitation visit 30 days after surgery
  Interventions: Drug: ferrous glycine sulphate

INTERVENTIONS:
Drug: Ferric carboxymaltose — Single intravenous dose ferric carboxymaltose
  Other Names: intravenous iron
  Arms: Ferric carboxymaltose
Drug: ferrous glycine sulphate — Daily oral dose of 100 mg iron (ferrous glycine sulphate)
  Other Names: Oral iron
  Arms: Ferrous glycine sulphate

SUMMARY:
Postoperative anaemia are common in patients undergoing major orthopaedic surgery. The main consequence of perioperative anaemia is an increased risk of red blood cell (RBC) transfusions. Allogeneic RBC transfusion and anaemia are associated with higher postoperative mortality and morbidity.

The aim of this study was to compare the efficacy of postoperative i.v. ferric carboxymaltose (FCM) and oral ferrous glycine sulphate (FS) for early improvement of postoperative anaemia after total knee arthroplasty and whether iron treatment could facilitate recovery from surgery.

DETAILED DESCRIPTION:
Both pre- and postoperative anaemia are common in patients undergoing major orthopaedic surgery. The main consequence of perioperative anaemia is an increased risk of red blood cell (RBC) transfusions. Allogeneic RBC transfusion and anaemia are associated with higher postoperative mortality and morbidity. Since blood transfusions increase Hb levels only transiently but come at the price of higher mortality and morbidity (e.g. postoperative infections), the three-pillar concept of patient blood management (PBM) has been developed to reduce the risk of blood transfusions and improve patient outcomes. Among its three pillars, the treatment or prevention of preoperative anaemia is the mainstay of PBM. Also the second pillar, minimisation of intraoperative blood loss,15 targets at least indirectly the patient's haemoglobin (Hb) levels.

The third PBM pillar, use of low Hb cut-off levels triggering transfusion, means that a certain degree of postoperative anaemia is taken into account. However, it remains unclear whether a lowered transfusion threshold allows optimal functional recovery and quality of life. Since patients undergoing total knee arthroplasty (TKA) are often elderly and have several comorbidities, prolonged exposure to low Hb levels is not a good option for this population. Furthermore, TKA patients should be mobilised as soon as possible after surgery which increases the metabolic demand.

Although, depending on the timescale before surgery, oral iron is suggested for preoperatively anaemic patients with absolute iron deficiency, oral iron showed no benefit over placebo in anaemic patients after lower limb arthroplasty. In patients at risk of functional iron deficiency due to chronic inflammation of different aetiologies, intravenous (i.v.) iron administration has proven its superiority over oral iron. Even in iron-deficient patients without established anaemia, i.v. iron improved physical performance and cardiac functional class. Thus, postoperative anaemia treatment with i.v. iron might not only reduce RBC requirements but also improve performance, rehabilitation and outcomes.

The aim of this study was to compare the efficacy of postoperative i.v. ferric carboxymaltose (FCM) and oral ferrous glycine sulphate (FS) for early improvement of postoperative anaemia after total knee arthroplasty and whether iron treatment could facilitate recovery from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age) were recruited at the scheduled preoperative visit (21 to 30 days prior surgery knee replacement). Anaemia (Hb <12 g/dL) and/or iron deficiency (TSAT <20%) the day after surgery

Exclusion Criteria:

* Patients with known hypersensitivity or contraindications to iron, liver insufficiency (aspartate aminotransferase or alanine aminotransferase >60 IU/L), bronchial asthma, presence of acute or chronic infection, severe heart disease, significant history of allergies (rash, etc.) or anti-anaemia treatment within 15 days prior to surgery were excluded from participation. Also pregnant or nursing women were excluded (negative pregnancy urine test within 7 days prior first study treatment or amenorrhoea for at least 12 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin concentration | 30 days
  Change in hemoglobin concentrations from baseline to 30 days

SECONDARY OUTCOMES:
Anemia | 30 days
  Number of subjects without anemia (hemoglobin > 12g/dL)
Hemoglobin concentration | 30 days
  Concentration of hemoglobin at day 30
Quality of life | 30 days
  Quality of life measured by European Quality of Life-5 Dimensions (EQ-5D)(before and 30 days)
Independence in daily activities | 30 days
  Independence in daily activities measured by the Barthel questionnaire (before and 30 days)
Walk test | 30 days
  6 minutes walking test (before and 30 days)
Adverse events | 30 days
  Adverse event (clinical and analytical, before to 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Bisbe, MD, Study Director — Parc de Salut Mar; Luis Molto, MD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Hospital de la Esperanza (Parc de Salut MAR), Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Bisbe E, Molto L, Arroyo R, Muniesa JM, Tejero M. Randomized trial comparing ferric carboxymaltose vs oral ferrous glycine sulphate for postoperative anaemia after total knee arthroplasty. Br J Anaesth. 2014 Sep;113(3):402-9. doi: 10.1093/bja/aeu092. Epub 2014 Apr 29. PMID 24780615